## THE EFFECT OF NURSING INTERVENTIONS BASED ON CONSERVATION MOTIVATION THEORY ON DRUG ADHERENCE AND HEALTHY LİFESTYLE BEHAVIORS İN PATIENTS WİTH HYPERTENSION: A RANDOMİZED CONTROLLED STUDY

NCT05995977

**Document Date: 20 June 2024** 

## Statistical Analysis Plan

In this study, data analysis was performed using the IBM SPSS Statistics Standard Concurrent User V 26 (IBM Corp., Armonk, New York, USA) program. Descriptive statistics were given as unit number (n), percentage (%), mean (X), standard deviation (SS), median (M), minimum (min) and maximum (max) values. Reliability for scales and their sub-dimensions was examined using Cronbach's Alpha coefficient. Scales with a Cronbach's Alpha coefficient above 0.60 were considered reliable. Skewness and kurtosis values were examined to test whether the data met the assumption of normality. In the decision stage, if the absolute skewness (Skewness) value is below  $\pm 2.0$  and the kurtosis value is below 7.0, it is decided that the data is normally distributed (Kim, 2013). Accordingly, the skewness and kurtosis values of the variables used in the study are given in Table 3.6 and it was found that the data were suitable for normal distribution. Independent sample t test was used to compare numerical descriptive characteristics of patients between groups, and chi-square tests (Pearson chi-square/Fisher exact test) were used to compare categorical descriptive characteristics between groups. Mixed order analysis of variance (ANOVA) was used to compare variables according to follow-up times in groups. Bonferroni correction was applied to compare main effects in the analyses. A p value of <0.05 was considered statistically significant.

Intention to treat (ITT) analysis was performed in the evaluation of the data. ITT is a basic method used in maintaining randomization and preventing bias in case of withdrawal from the study. The approach to be applied when handling missing data varies according to whether the data is discrete or continuous. The most common method used in filling in missing data in continuous data is to fill in the last observed data by repeating the outcome measurements (Last Observation Carried Forward). Since it was not possible to reach 7 individuals who dropped out during the research process for the ITT analysis of this study, the post-tests were filled in by repeating the answers given by the patients in the pre-tests and the missing data were completed in this way. A summary of the statistics used in this study is shown in Table 1.

Table 1. Statistics used in the study (n=78).

| Evaluated statistics | Statistical methods |
|---|---|
| Normal distribution | Skewness and kurtosis values |
| In comparing numerical descriptive characteristics between groups | Independent Sample t Test |
| In comparing categorical descriptive characteristics between groups | From chi-square tests (Pearson chi-square/Fisher exact test) |
| In comparing variables in groups according to follow-up times | Mixed order analysis of variance (ANOVA) |
| In comparing main effects in analyses | Bonferroni correction |
| Reliability for scales and their sub-<br>dimensions | Cronbach's Alpha coefficient |
| In evaluating missing data | intention to treat (ITT) analysis |